CLINICAL TRIAL: NCT06957054
Title: Assessment of Neural Biomarkers in Adult Subjects With Fragile X Syndrome and Typically Developing Subjects
Brief Title: Neural Biomarkers in Fragile X Syndrome
Acronym: EXP-CTH120
Status: Completed | Type: Observational
Sponsor: Connecta Therapeutics, S.L. (Industry)
Collaborators: Hospital del Mar Research Institute (IMIM) (Other); Corporacion Parc Tauli (Other); Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Sponsor
Other Study IDs: CTH-CTH120-EXP-01
Record Dates: First submitted 2025-04-10; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Fragile X Syndrome (FXS); Neurotypical Adults
Keywords: Fragile X Syndrome; FXS; Fragile X; Neurodevelopmental Disorders; Central Nervous System Diseases; Intellectual Disability; Neurobehavioral Manifestations; Genetic Diseases, X-Linked; Congenital Abnormalities; Orphan Diseases; Rare Diseases; Neural biomarkers
MeSH Terms: conditions — Fragile X Syndrome; Neurodevelopmental Disorders; Central Nervous System Diseases; Intellectual Disability; Neurobehavioral Manifestations; Genetic Diseases, X-Linked; Congenital Abnormalities; Rare Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, urine and hair samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Fragile X syndrome
  Interventions: Other: Any
- Group 2: Typically Developing Subjects
  Interventions: Other: Any

INTERVENTIONS:
Other: Any — Any

SUMMARY:
The purpose of this non-interventional test /re-test study is to assess neural biomarkers in adult subjects with Fragile X syndrome compared to those measured in a population of typically developing adults

DETAILED DESCRIPTION:
This study consists of a screening period and two cross sectional evaluations assessed in one month interval (test/re-test), first on the Visit 1 (Basal) and the other on the Visit 2 (end-of-study visit, EOS).

ELIGIBILITY:
Demographics common to all subjects:

* Male or female subjects.
* Age ≥ 18 and ≤ 55 years.
* Weight ≥ 50 kg and ≤ 100 kg.
* Body mass index (BMI) ≥ 18.5 and ≤ 30.

Subjects with Fragile X syndrome Inclusion Criteria:

* Clinical and molecular diagnosis of Fragile X syndrome (> 200 CGG repeats in the promoter region of the FMR1 gene).
* Legal representative understands and accepts the study procedures. If only one parent signs, he/she should confirm that the other parent does not object to the patient's participation in the research project.
* Subject assenting and/or willing to participate.
* Signed informed consent by a legal representative before any study-mandated procedure.
* Subject is independently mobile and has sufficient vision and hearing to participate in study evaluations. They must be able to be understood most of the time and must not use other forms of communication, signs, symbol boards or devices as their primary form of communication.
* Subjects must have a parent, or other reliable caregiver, who agrees to accompany the subject to all study visits, provide information about the subject as required by the protocol, and ensure compliance with study tests.
* Subjects are expected to complete all procedures scheduled during the study visits.

Subjects with Fragile X syndrome Exclusion Criteria:

* Personal history of infantile spasms/convulsions/epilepsy, severe head trauma or CNS infections (e.g. meningitis), with the exception of infantile febrile seizures.
* Subjects with a current diagnosis including severe autism spectrum disorder or any primary psychiatric diagnosis according to DSM-5 (Diagnostic and Statistical Manual of Mental Disorders-DSM-5). Diagnoses that are secondary, such as attention deficit hyperactivity disorder, depressive disorders and conduct disorders are allowed as long as they are considered to not interfere with study conduct and are stable during the 3 months before inclusion. Related allowed treatments must be on stable dosing for the last 3 months.
* Substance use disorder according to the DSM-5 criteria.
* Epileptiform abnormalities (excluding isolated sharp waves and beyond those expected for age).
* Any life-threatening disease.
* Any other clinically relevant concomitant disease or condition or finding at screening that in the judgment of the investigator could interfere with, the treatment thereof might interfere with, the conduct of the study and related procedures and/or might bias the study results interpretation, or could jeopardize the subject's safety.
* Any clinically significant findings in physical examination including vital signs.
* Neuroleptic or antidepressant (ISRS) drugs within 3 months before inclusion, except for sertraline at a maximum 100 mg/day, and stable for the last 3 months before inclusion.
* Any prescription or over-the-counter drug (except occasional use of paracetamol) in the last 2 weeks before screening.
* Patient included in a clinical study with drugs in the last three months prior to inclusion.

Typically Developing Subjects Inclusion Criteria:

* Abstinence for any drug abuse 72 hours prior to the screening visit and the observation days, except for nicotine (24 hours).
* Able to read Spanish and/or Catalan and to adhere to the study requirements.
* Signed informed consent prior to any study-mandated procedure.

Typically Developing Subjects Exclusion Criteria:

* Life-time clinically significant cardiovascular, renal, pulmonary, hepatic, onco-haematological, endocrine, gastrointestinal, mental or neurological disease.
* Any other clinically relevant concomitant disease or condition or finding at screening that in the judgment of the investigator could interfere with, the treatment thereof might interfere with, the conduct of the study and related procedures and/or might bias the study results interpretation, or could jeopardize the subject's safety.
* Any clinically significant findings in physical examination including vital signs.
* Neuroleptic drugs within 3 months prior to inclusion.
* Any prescription or over-the-counter drug (except occasional use of paracetamol) in the last 2 weeks before screening.
* Patient included in a clinical study with drugs in the last three months before inclusion.
* Personal history of infantile spasms/convulsions/epilepsy, severe head trauma or CNS infections (e.g. meningitis), except for infantile febrile seizures.
* Subjects with a current diagnosis including autism spectrum disorder or any primary psychiatric diagnosis according to DSM-5 (Diagnostic and Statistical Manual of Mental Disorders-DSM-5). Diagnoses that are secondary, such as attention deficit hyperactivity disorder, depressive disorders and conduct disorders are allowed as long as they are considered to not interfere with study conduct and are stable during the 3 months before inclusion. Related allowed treatments must be on stable dosing for the last 3 months.
* Substance use disorder according to the DSM-5 criteria except for mild alcohol use disorder and/or mild or moderate nicotine use disorder.
* Positive urine test for drugs of abuse or alcohol breath test at screening.
* Epileptiform abnormalities (excluding isolated sharp waves and beyond those expected for age).
* Any life-threatening disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fragile X syndrome adult patients compared to neurotypical adults
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Cognitive profile of FXS patients compared to neurotypical subjects using the NIH-TCB-ID Toolbox | Day 1 and Day 28 (± 3 days)
  The NIH-Toolbox Cognitive Battery for Intellectual Disabilities (NIH-TCB-ID) provides a reliable, validated and standardized measure (composite scores) that can be used as efficacy endpoints in clinical studies in patients with neurodevelopmental disorders from 3 to 85 years old. The Fluid Cognition composite score of the NIH Toolbox cognitive battery combines the scores of five tests assessing the following cognitive domains: i) Cognitive flexibility, ii) Inhibitory control and visual attention, iii) Episodic memory, iv) Processing speed and v) Working memory.
Neural oscillations using Electroencephalography (EEG) | Day 1
  Multichannel EEG will be recorded using a mobile wireless helmet for high precision EEG monitoring. In total, 20 EEG channels will be used to capture brainwave activity.
  The EEG test contains three well differentiated sections: auditory oddball, resting-state (eyes open and eyes closed) and auditory steady-state response (ASSR). Before starting the auditory oddball, the subject will conduct a training section (40 seconds) to present the type of sounds and to check that they have understood the task by practicing it.
Point of gaze using eye tracking | Day 1 and Day 28 (± 3 days)
  Eye tracking technology will be used to record X and Y coordinates of eye position and pupil diameter. Stimuli will consist on 60 coloured photographs of adult human faces (equal numbers of males and females; different races and ethnicities), each face exhibiting a calm, happy, or fearful expression, and 60 scrambled versions of the face images. Testing will be conducted in a quiet room with the lights turned off. Each trial will start with presentation of a scrambled face image for 1 s followed immediately by its matched face image for 3 s. An inter-trial interval (ITI) containing a uniform grey screen will be shown for 0.5, 1, or 2 s, randomly determined. The order of face presentation will be pseudorandomized and each eye tracking session will last approximately 6 min.
Behavior troubles of the FXS patients compared to neurotypical subjects using the Aberrant Behavior Checklist (ABC) | ≤ 1 month prior to Day 1
  Standardized rating scale used for assessing problematic behavior of individuals with developmental disabilities. The questionnaire explores problem behaviors across 5 domains: Irritability (15 items), Lethargy/Socially Withdrawal (16 items), Stereotypy Behavior (7 items), Hyperactivity/Noncompliance (16 items), Inappropriate Speech (4 items). Each item is scored as 0 (never a problem), 1 (slight problem), 2 (moderately serious problem), or 3 (severe problem). For the present study the total score for each of the 5 domains or subscales will be calculated and used for the analyses, as a good measure of the psychiatric symptom and behavioral disturbance profile. In all cases, higher scores in the mentioned subscales and total score indicated a greater presence and severity of behavioral problems: Agitation [0-45]; Lethargy/Social Withdrawal [0-48]; Stereotypic Behavior [0-21]; Hyperactivity/Noncompliance [0-48] and Inappropriate Speech [0-12].
Adaptative functioning using the Vineland Adaptive Behaviour Scale (VABS-3) | ≤ 1 month prior to Day 1
  The Vineland Adaptative Behaviour Scale 3 (VABS-3) is a psychometric instrument used in child and adolescent clinical psychology for the assessment of individuals with different types of developmental delays, regarding an adaptive level of functioning by standardized interview of the person or their caregiver through their activities of daily living such as walking, talking, getting dressed, going to school, preparing a meal, etc. Three domains explore communication, socialization and daily living, which correspond to the 3 domains of adaptive functioning recognized by the American Association on Intellectual and Developmental Disabilities.
Clinician-rated global functioning using the Clinical Global Impression (CGI) | ≤ 1 month prior to Day 1 and Day 28 (± 3 days)
  The Clinical Global Impression Scale (CGI) comprises two companion one-item measures evaluating the following:
  1. Severity of Psychopathology (Clinical Global Impression-Severity (CGI-S) Scale): establishes the baseline illness status and rates illness severity on a 7-point scale [range 0 to 7]: 1 for not at all ill; 2 for borderline illness; 3 for mild illness; 4 for moderately ill; 5 for very ill; 6 for severely ill; 7 among the most severe patients; and
  2. Change from the Initiation of Treatment (Clinical Global Impression-Improvement (CGI-I) Scale): rates how much the subject's illness has improved or worsened relative to the baseline state (CGI-S) on a 7-point scale [range -7 to 7]: 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; and 7 = very much worse.
Stress biomarkers of the FXS patients compared to neurotypical subjects measured by cortisol concentrations in hair (occipital area) | ≤ 1 month prior to Day 1
  Hair cortisol analysis characterizes chronic stress as a risk factor for chronic illness progression and is known as a biomarker of the effectiveness of stress reduction interventions. Approximately 3 cm of occipital hair will be collected at the Screening visit for the determination of cortisol concentrations [range 2.5 - 97.5 pg/mg].
Biorhythm characteristics of FXS patients compared to neurotypical subjects determining vitamin D (25-Hydroxy) concentrations in serum | Day 1 and Day 28 (± 3 days)
  Vitamin D concentrations are also useful due to lack of sunlight exposure is the primary reason for the worldwide epidemic of vitamin D deficiency. The lack of sunlight exposure is involved in serotonin and melatonin production. Venous blood samples will be collected by individual venepuncture or via an indwelling catheter to measure vitamin D (25-Hydroxy) concentrations in serum [25 - 150 ng/mL].
Biorhythm characteristics of FXS patients compared to neurotypical subjects determining 24h urine cortisol concentrations | Day 1 and Day 28 (± 3 days)
  The activation of the Hypothalamic Pituitary Adrenal (HPA) axis leads to the synthesis and release of cortisol, a glucocorticoid hormone that peaks in the early morning hours. 24-hour urine samples will be collected before Visit 1 and Visit 2 for the determination of cortisol concentrations [range 11.5 - 102.0 µg/24h].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using sleep diaries | From Day 1 to Day 28 (± 3 days)
  Sleep schedule will be assessed by using sleep diaries to record the quality and quantity of sleep. A sleep diary allows recording when the subject goes to bed, when the subject wakes up during the night and when the subject wakes up in the morning. This will help to understand the sleep pattern and how much sleep the subject gets. It will also show how often the subject has interrupted sleep.
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: number of days | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the number of days [days].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: percentage of wear | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the percentage of wear [%].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: total steps | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the total steps [steps].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: steps per day | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the steps per day [steps/day].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: average of energy expenditure | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the average of energy expenditure [kcal/day].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: percentage of sedentary physical activity | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the percentage of sedentary physical activity [%].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: percentage of light physical activity | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the percentage of light physical activity [%].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: percentage of moderate physical activity | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the percentage of moderate physical activity [%].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: percentage of vigorous physical activity | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the percentage of vigorous physical activity [%].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: percentage of very vigorous physical activity | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the percentage of very vigorous physical activity [%].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: bedtime | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the bedtime [hh:mm].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: wake-up time | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the wake-up time [hh:mm].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: mean time in bed | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the mean time in bed [minutes].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: total mean sleep time | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the total mean sleep time [minutes].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: sleep efficiency | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the sleep efficiency [%].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: wake after sleep onset | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the wake after sleep onset [minutes].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: average of awakening | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the average of awakening [awakes].
Biorhythm characteristics of FXS patients compared to neurotypical subjects using actigraphy: hours spent awake at night | From Day 1 to Day 28 (± 3 days)
  Sleep-wake rhythms will be assessed using a wearable actigraph which will register the hours spent awake at night [minutes].
Quality of life of the FXS patients compared to neurotypical subjects using the Paediatric Quality of Life Inventory (PedsQL) | ≤ 1 month prior to Day 1
  Health-related quality of life (HRQoL) is a multidimensional concept involving physical, psychological, social, and cognitive aspects of life. Individuals with Fragile X syndrome (FXS) experience a life-long disorder that impacts the HRQoL of the affected individual and their family. HRQoL has been correlated with established measures of functioning in FXS using the: i) Cognitive Functioning Scale [0-100], ii) Quality of Life Scale, which is composite of the following items: Physical health and activities [0-32], Emotional state [0-20], Social activities [range 0-20], School activities [0-20]; and iii) Family impact scale, which is composite of the following items: Physical health and activities [0-24], Emotional state [0-20], Social activities [0-16], Cognitive function [0-20], Communication [0-12], Preoccupation [0-20], Daily activities [0-12] and Family relationships [0-20].
Quality of sleep of the FXS patients compared to neurotypical subjects using Pittsburgh sleep quality index (PSQI) | Day 1 and Day 28 (± 3 days)
  The Pittsburgh sleep quality index (PSQI) consists in a self-report questionnaire that assesses sleep quality and quantity. The 19-item self-report questionnaire yields 7 component scores: i) subjective sleep quality [0-3], ii) sleep latency [0-3], ii) duration of the sleep [0-3], iii) habitual sleep efficiency [0-3], iv) sleep disturbances [0-3], v) use of sleeping medication [0-3], and vi) daytime dysfunction [0-3]. There are five additional questions that are completed by a bed partner if there is one.
FMRP protein in peripheral blood of FXS patients in peripheral blood compared to neurotypical subjects | ≤ 1 month prior to Day 1
  Venous blood samples will be obtained by extraction of peripheral blood from participants in a EDTA tube. The levels of FMRP in the FMR1 gene will be reported as a relative value of the mean levels calculated for control [range 0-1].
miRNA profile of FXS patients in plasma compared to neurotypical subjects | Day 1 and Day 28 (± 3 days)
  Venous blood samples will be obtained by extraction of peripheral blood from participants. For the determination of the miRNomic profile, 200 μL of human plasma will be processed using Plasma/Serum miRNeasy Serum/Plasma kit to extract RNA enriched in small RNAs.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael De la Torre Fornell, Pharm, PhD, Principal Investigator — Hospital del Mar Research Institute; Ana Roche Martínez, MD, PhD, Principal Investigator — Consorci Corporació Sanitària Parc Taulí. Institut d'Investigació i Innovació Parc Taulí (I3PT)
Locations (2):
- Spain (2):
  - Hospital del Mar Research Institute (HMRI), Barcelona, Barcelona
  - Consorci Corporació Sanitaria Parc Taulí. Institut Investigació i Innovació Parc Taulí (I3PT), Sabadell, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sotoudeh Anvari M, Vasei H, Najmabadi H, Badv RS, Golipour A, Mohammadi-Yeganeh S, Salehi S, Mohamadi M, Goodarzynejad H, Mowla SJ. Identification of microRNAs associated with human fragile X syndrome using next-generation sequencing. Sci Rep. 2022 Mar 23;12(1):5011. doi: 10.1038/s41598-022-08916-4. PMID 35322102
- [Background] Couto RR, Kubaski F, Siebert M, Felix TM, Brusius-Facchin AC, Leistner-Segal S. Increased Serum Levels of miR-125b and miR-132 in Fragile X Syndrome: A Preliminary Study. Neurol Genet. 2022 Oct 26;8(6):e200024. doi: 10.1212/NXG.0000000000200024. eCollection 2022 Dec. PMID 36313066
- [Background] Lin SL. microRNAs and Fragile X Syndrome. Adv Exp Med Biol. 2015;888:107-21. doi: 10.1007/978-3-319-22671-2_7. PMID 26663181
- [Background] Daly I, Pichiorri F, Faller J, Kaiser V, Kreilinger A, Scherer R, Muller-Putz G. What does clean EEG look like? Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:3963-6. doi: 10.1109/EMBC.2012.6346834. PMID 23366795
- [Background] Castren M, Paakkonen A, Tarkka IM, Ryynanen M, Partanen J. Augmentation of auditory N1 in children with fragile X syndrome. Brain Topogr. 2003 Spring;15(3):165-71. doi: 10.1023/a:1022606200636. PMID 12705812
- [Background] Kenny A, Wright D, Stanfield AC. EEG as a translational biomarker and outcome measure in fragile X syndrome. Transl Psychiatry. 2022 Jan 24;12(1):34. doi: 10.1038/s41398-022-01796-2. PMID 35075104
- [Background] Varni JW, Limbers CA. The PedsQL 4.0 Generic Core Scales Young Adult Version: feasibility, reliability and validity in a university student population. J Health Psychol. 2009 May;14(4):611-22. doi: 10.1177/1359105309103580. PMID 19383661
- [Background] Aman MG, Norris M, Kaat AJ, Andrews H, Choo TH, Chen C, Wheeler A, Bann C, Erickson C. Factor Structure of the Aberrant Behavior Checklist in Individuals with Fragile X Syndrome: Clarifications and Future Guidance. J Child Adolesc Psychopharmacol. 2020 Oct;30(8):512-521. doi: 10.1089/cap.2019.0177. Epub 2020 Aug 3. PMID 32746626
- [Background] Prosser H, Moss S, Costello H, Simpson N, Patel P, Rowe S. Reliability and validity of the Mini PAS-ADD for assessing psychiatric disorders in adults with intellectual disability. J Intellect Disabil Res. 1998 Aug;42 ( Pt 4):264-72. doi: 10.1046/j.1365-2788.1998.00146.x. PMID 9786440
- [Background] Shields RH, Kaat AJ, McKenzie FJ, Drayton A, Sansone SM, Coleman J, Michalak C, Riley K, Berry-Kravis E, Gershon RC, Widaman KF, Hessl D. Validation of the NIH Toolbox Cognitive Battery in intellectual disability. Neurology. 2020 Mar 24;94(12):e1229-e1240. doi: 10.1212/WNL.0000000000009131. Epub 2020 Feb 24. PMID 32094241
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Tottenham N, Tanaka JW, Leon AC, McCarry T, Nurse M, Hare TA, Marcus DJ, Westerlund A, Casey BJ, Nelson C. The NimStim set of facial expressions: judgments from untrained research participants. Psychiatry Res. 2009 Aug 15;168(3):242-9. doi: 10.1016/j.psychres.2008.05.006. Epub 2009 Jun 28. PMID 19564050
- [Background] Bailey DB Jr, Berry-Kravis E, Wheeler A, Raspa M, Merrien F, Ricart J, Koumaras B, Rosenkranz G, Tomlinson M, von Raison F, Apostol G. Mavoglurant in adolescents with fragile X syndrome: analysis of Clinical Global Impression-Improvement source data from a double-blind therapeutic study followed by an open-label, long-term extension study. J Neurodev Disord. 2016;8:1. doi: 10.1186/s11689-015-9134-5. Epub 2015 Dec 15. PMID 26855682
- [Background] Tassone F, Hagerman RJ, Taylor AK, Gane LW, Godfrey TE, Hagerman PJ. Elevated levels of FMR1 mRNA in carrier males: a new mechanism of involvement in the fragile-X syndrome. Am J Hum Genet. 2000 Jan;66(1):6-15. doi: 10.1086/302720. PMID 10631132
- [Background] Zafarullah M, Li J, Salemi MR, Phinney BS, Durbin-Johnson BP, Hagerman R, Hessl D, Rivera SM, Tassone F. Blood Proteome Profiling Reveals Biomarkers and Pathway Alterations in Fragile X PM at Risk for Developing FXTAS. Int J Mol Sci. 2023 Aug 30;24(17):13477. doi: 10.3390/ijms241713477. PMID 37686279
- [Background] Bowling H, Bhattacharya A, Zhang G, Alam D, Lebowitz JZ, Bohm-Levine N, Lin D, Singha P, Mamcarz M, Puckett R, Zhou L, Aryal S, Sharp K, Kirshenbaum K, Berry-Kravis E, Neubert TA, Klann E. Altered steady state and activity-dependent de novo protein expression in fragile X syndrome. Nat Commun. 2019 Apr 12;10(1):1710. doi: 10.1038/s41467-019-09553-8. PMID 30979884
- [Background] AlOlaby RR, Sweha SR, Silva M, Durbin-Johnson B, Yrigollen CM, Pretto D, Hagerman RJ, Tassone F. Molecular biomarkers predictive of sertraline treatment response in young children with fragile X syndrome. Brain Dev. 2017 Jun;39(6):483-492. doi: 10.1016/j.braindev.2017.01.012. Epub 2017 Feb 24. PMID 28242040
- [Background] Bekheet MHY, Mansour LA, Elkaffas RH, Kamel MA, Elmonem MA. Serum matrix metalloproteinase-9 (MMP9) and amyloid-beta protein precursor (APP) as potential biomarkers in children with Fragile-X syndrome: A cross sectional study. Clin Biochem. 2023 Nov;121-122:110659. doi: 10.1016/j.clinbiochem.2023.110659. Epub 2023 Oct 4. PMID 37797798
- [Background] Dionne O, Corbin F. A new strategy to uncover fragile X proteomic biomarkers using the nascent proteome of peripheral blood mononuclear cells (PBMCs). Sci Rep. 2021 Jul 26;11(1):15148. doi: 10.1038/s41598-021-94027-5. PMID 34312401
- [Background] Zafarullah M, Tassone F. Molecular Biomarkers in Fragile X Syndrome. Brain Sci. 2019 Apr 27;9(5):96. doi: 10.3390/brainsci9050096. PMID 31035599
- [Background] Hessl D, Glaser B, Dyer-Friedman J, Blasey C, Hastie T, Gunnar M, Reiss AL. Cortisol and behavior in fragile X syndrome. Psychoneuroendocrinology. 2002 Oct;27(7):855-72. doi: 10.1016/s0306-4530(01)00087-7. PMID 12183220
- [Background] Russell E, Koren G, Rieder M, Van Uum S. Hair cortisol as a biological marker of chronic stress: current status, future directions and unanswered questions. Psychoneuroendocrinology. 2012 May;37(5):589-601. doi: 10.1016/j.psyneuen.2011.09.009. Epub 2011 Oct 4. PMID 21974976
- [Background] Wright KD, Hickman R, Laudenslager ML. Hair Cortisol Analysis: A Promising Biomarker of HPA Activation in Older Adults. Gerontologist. 2015 Jun;55 Suppl 1(Suppl 1):S140-5. doi: 10.1093/geront/gnu174. PMID 26055775
- [Background] Prono F, Bernardi K, Ferri R, Bruni O. The Role of Vitamin D in Sleep Disorders of Children and Adolescents: A Systematic Review. Int J Mol Sci. 2022 Jan 27;23(3):1430. doi: 10.3390/ijms23031430. PMID 35163353
- [Background] Hardiman RL, Bratt A. Hypothalamic-pituitary-adrenal axis function in Fragile X Syndrome and its relationship to behaviour: A systematic review. Physiol Behav. 2016 Dec 1;167:341-353. doi: 10.1016/j.physbeh.2016.09.030. Epub 2016 Oct 5. PMID 27720735
- [Background] Dueck A, Reis O, Bastian M, van Treeck L, Weirich S, Haessler F, Fiedler A, Koelch M, Berger C. Feasibility of a Complex Setting for Assessing Sleep and Circadian Rhythmicity in a Fragile X Cohort. Front Psychiatry. 2020 May 14;11:361. doi: 10.3389/fpsyt.2020.00361. eCollection 2020. PMID 32477175
- [Background] Farzin F, Scaggs F, Hervey C, Berry-Kravis E, Hessl D. Reliability of eye tracking and pupillometry measures in individuals with fragile X syndrome. J Autism Dev Disord. 2011 Nov;41(11):1515-22. doi: 10.1007/s10803-011-1176-2. PMID 21267642
- [Background] Klusek J, Moser C, Schmidt J, Abbeduto L, Roberts JE. A novel eye-tracking paradigm for indexing social avoidance-related behavior in fragile X syndrome. Am J Med Genet B Neuropsychiatr Genet. 2020 Jan;183(1):5-16. doi: 10.1002/ajmg.b.32757. Epub 2019 Aug 16. PMID 31418535
- [Background] Ethridge LE, Pedapati EV, Schmitt LM, Norris JE, Auger E, De Stefano LA, Sweeney JA, Erickson CA. Validating brain activity measures as reliable indicators of individual diagnostic group and genetically mediated sub-group membership Fragile X Syndrome. Res Sq [Preprint]. 2024 Jan 18:rs.3.rs-3849272. doi: 10.21203/rs.3.rs-3849272/v1. PMID 38313274
- [Background] Coffee B, Keith K, Albizua I, Malone T, Mowrey J, Sherman SL, Warren ST. Incidence of fragile X syndrome by newborn screening for methylated FMR1 DNA. Am J Hum Genet. 2009 Oct;85(4):503-14. doi: 10.1016/j.ajhg.2009.09.007. PMID 19804849
- [Background] Hunter J, Rivero-Arias O, Angelov A, Kim E, Fotheringham I, Leal J. Epidemiology of fragile X syndrome: a systematic review and meta-analysis. Am J Med Genet A. 2014 Jul;164A(7):1648-58. doi: 10.1002/ajmg.a.36511. Epub 2014 Apr 3. PMID 24700618
- [Background] Tassone F, Iong KP, Tong TH, Lo J, Gane LW, Berry-Kravis E, Nguyen D, Mu LY, Laffin J, Bailey DB, Hagerman RJ. FMR1 CGG allele size and prevalence ascertained through newborn screening in the United States. Genome Med. 2012 Dec 21;4(12):100. doi: 10.1186/gm401. eCollection 2012. PMID 23259642
- [Background] Crawford DC, Acuna JM, Sherman SL. FMR1 and the fragile X syndrome: human genome epidemiology review. Genet Med. 2001 Sep-Oct;3(5):359-71. doi: 10.1097/00125817-200109000-00006. PMID 11545690
- [Background] Kidd SA, Lachiewicz A, Barbouth D, Blitz RK, Delahunty C, McBrien D, Visootsak J, Berry-Kravis E. Fragile X syndrome: a review of associated medical problems. Pediatrics. 2014 Nov;134(5):995-1005. doi: 10.1542/peds.2013-4301. Epub 2014 Oct 6. PMID 25287458
- [Background] Rajan-Babu IS, Chong SS. Molecular Correlates and Recent Advancements in the Diagnosis and Screening of FMR1-Related Disorders. Genes (Basel). 2016 Oct 14;7(10):87. doi: 10.3390/genes7100087. PMID 27754417
- [Background] Tassone F. Advanced technologies for the molecular diagnosis of fragile X syndrome. Expert Rev Mol Diagn. 2015;15(11):1465-73. doi: 10.1586/14737159.2015.1101348. Epub 2015 Oct 21. PMID 26489042
- [Background] Leehey MA. Fragile X-associated tremor/ataxia syndrome: clinical phenotype, diagnosis, and treatment. J Investig Med. 2009 Dec;57(8):830-6. doi: 10.2310/JIM.0b013e3181af59c4. PMID 19574929
- [Background] Utari A, Adams E, Berry-Kravis E, Chavez A, Scaggs F, Ngotran L, Boyd A, Hessl D, Gane LW, Tassone F, Tartaglia N, Leehey MA, Hagerman RJ. Aging in fragile X syndrome. J Neurodev Disord. 2010 Jun;2(2):70-76. doi: 10.1007/s11689-010-9047-2. Epub 2010 May 12. PMID 20585378
- [Background] Cordeiro L, Ballinger E, Hagerman R, Hessl D. Clinical assessment of DSM-IV anxiety disorders in fragile X syndrome: prevalence and characterization. J Neurodev Disord. 2011 Mar;3(1):57-67. doi: 10.1007/s11689-010-9067-y. Epub 2010 Dec 3. PMID 21475730
- [Background] Bartholomay KL, Lee CH, Bruno JL, Lightbody AA, Reiss AL. Closing the Gender Gap in Fragile X Syndrome: Review on Females with FXS and Preliminary Research Findings. Brain Sci. 2019 Jan 12;9(1):11. doi: 10.3390/brainsci9010011. PMID 30642066
- [Background] Sauna-Aho O, Bjelogrlic-Laakso N, Siren A, Arvio M. Signs indicating dementia in Down, Williams and Fragile X syndromes. Mol Genet Genomic Med. 2018 Sep;6(5):855-860. doi: 10.1002/mgg3.430. Epub 2018 Jul 3. PMID 29971948
- [Background] McLennan Y, Polussa J, Tassone F, Hagerman R. Fragile x syndrome. Curr Genomics. 2011 May;12(3):216-24. doi: 10.2174/138920211795677886. PMID 22043169
- [Background] Bailey DB Jr, Raspa M, Olmsted M, Holiday DB. Co-occurring conditions associated with FMR1 gene variations: findings from a national parent survey. Am J Med Genet A. 2008 Aug 15;146A(16):2060-9. doi: 10.1002/ajmg.a.32439. PMID 18570292
- [Background] Pilaz LJ, Lennox AL, Rouanet JP, Silver DL. Dynamic mRNA Transport and Local Translation in Radial Glial Progenitors of the Developing Brain. Curr Biol. 2016 Dec 19;26(24):3383-3392. doi: 10.1016/j.cub.2016.10.040. Epub 2016 Dec 1. PMID 27916527
- [Background] Danesi C, Achuta VS, Corcoran P, Peteri UK, Turconi G, Matsui N, Albayrak I, Rezov V, Isaksson A, Castren ML. Increased Calcium Influx through L-type Calcium Channels in Human and Mouse Neural Progenitors Lacking Fragile X Mental Retardation Protein. Stem Cell Reports. 2018 Dec 11;11(6):1449-1461. doi: 10.1016/j.stemcr.2018.11.003. Epub 2018 Nov 29. PMID 30503263
- [Background] Pasciuto E, Ahmed T, Wahle T, Gardoni F, D'Andrea L, Pacini L, Jacquemont S, Tassone F, Balschun D, Dotti CG, Callaerts-Vegh Z, D'Hooge R, Muller UC, Di Luca M, De Strooper B, Bagni C. Dysregulated ADAM10-Mediated Processing of APP during a Critical Time Window Leads to Synaptic Deficits in Fragile X Syndrome. Neuron. 2015 Jul 15;87(2):382-98. doi: 10.1016/j.neuron.2015.06.032. PMID 26182420
- [Background] Sidhu H, Dansie LE, Hickmott PW, Ethell DW, Ethell IM. Genetic removal of matrix metalloproteinase 9 rescues the symptoms of fragile X syndrome in a mouse model. J Neurosci. 2014 Jul 23;34(30):9867-79. doi: 10.1523/JNEUROSCI.1162-14.2014. PMID 25057190
- [Background] Kashima R, Roy S, Ascano M, Martinez-Cerdeno V, Ariza-Torres J, Kim S, Louie J, Lu Y, Leyton P, Bloch KD, Kornberg TB, Hagerman PJ, Hagerman R, Lagna G, Hata A. Augmented noncanonical BMP type II receptor signaling mediates the synaptic abnormality of fragile X syndrome. Sci Signal. 2016 Jun 7;9(431):ra58. doi: 10.1126/scisignal.aaf6060. PMID 27273096
- [Background] Wahlstrom-Helgren S, Klyachko VA. GABAB receptor-mediated feed-forward circuit dysfunction in the mouse model of fragile X syndrome. J Physiol. 2015 Nov 15;593(22):5009-24. doi: 10.1113/JP271190. Epub 2015 Oct 2. PMID 26282581
- [Background] Gkogkas CG, Khoutorsky A, Cao R, Jafarnejad SM, Prager-Khoutorsky M, Giannakas N, Kaminari A, Fragkouli A, Nader K, Price TJ, Konicek BW, Graff JR, Tzinia AK, Lacaille JC, Sonenberg N. Pharmacogenetic inhibition of eIF4E-dependent Mmp9 mRNA translation reverses fragile X syndrome-like phenotypes. Cell Rep. 2014 Dec 11;9(5):1742-1755. doi: 10.1016/j.celrep.2014.10.064. Epub 2014 Nov 26. PMID 25466251
- [Background] Wang H, Wu LJ, Kim SS, Lee FJ, Gong B, Toyoda H, Ren M, Shang YZ, Xu H, Liu F, Zhao MG, Zhuo M. FMRP acts as a key messenger for dopamine modulation in the forebrain. Neuron. 2008 Aug 28;59(4):634-47. doi: 10.1016/j.neuron.2008.06.027. PMID 18760699
- [Background] Chandana SR, Behen ME, Juhasz C, Muzik O, Rothermel RD, Mangner TJ, Chakraborty PK, Chugani HT, Chugani DC. Significance of abnormalities in developmental trajectory and asymmetry of cortical serotonin synthesis in autism. Int J Dev Neurosci. 2005 Apr-May;23(2-3):171-82. doi: 10.1016/j.ijdevneu.2004.08.002. PMID 15749243
- [Background] Boccuto L, Chen CF, Pittman AR, Skinner CD, McCartney HJ, Jones K, Bochner BR, Stevenson RE, Schwartz CE. Decreased tryptophan metabolism in patients with autism spectrum disorders. Mol Autism. 2013 Jun 3;4(1):16. doi: 10.1186/2040-2392-4-16. PMID 23731516
- [Background] Hanson AC, Hagerman RJ. Serotonin dysregulation in Fragile X Syndrome: implications for treatment. Intractable Rare Dis Res. 2014 Nov;3(4):110-7. doi: 10.5582/irdr.2014.01027. PMID 25606361
- [Background] Feng Y, Gutekunst CA, Eberhart DE, Yi H, Warren ST, Hersch SM. Fragile X mental retardation protein: nucleocytoplasmic shuttling and association with somatodendritic ribosomes. J Neurosci. 1997 Mar 1;17(5):1539-47. doi: 10.1523/JNEUROSCI.17-05-01539.1997. PMID 9030614
- [Background] Gholizadeh S, Halder SK, Hampson DR. Expression of fragile X mental retardation protein in neurons and glia of the developing and adult mouse brain. Brain Res. 2015 Jan 30;1596:22-30. doi: 10.1016/j.brainres.2014.11.023. Epub 2014 Nov 20. PMID 25446451
- [Background] Richter JD, Bassell GJ, Klann E. Dysregulation and restoration of translational homeostasis in fragile X syndrome. Nat Rev Neurosci. 2015 Oct;16(10):595-605. doi: 10.1038/nrn4001. Epub 2015 Sep 9. PMID 26350240
- [Background] Darnell JC, Klann E. The translation of translational control by FMRP: therapeutic targets for FXS. Nat Neurosci. 2013 Nov;16(11):1530-6. doi: 10.1038/nn.3379. Epub 2013 Apr 14. PMID 23584741
- [Background] Bakker CE, Oostra BA. Understanding fragile X syndrome: insights from animal models. Cytogenet Genome Res. 2003;100(1-4):111-23. doi: 10.1159/000072845. PMID 14526171
- [Background] Banerjee A, Ifrim MF, Valdez AN, Raj N, Bassell GJ. Aberrant RNA translation in fragile X syndrome: From FMRP mechanisms to emerging therapeutic strategies. Brain Res. 2018 Aug 15;1693(Pt A):24-36. doi: 10.1016/j.brainres.2018.04.008. Epub 2018 Apr 10. PMID 29653083
- [Background] Grigsby J. The fragile X mental retardation 1 gene (FMR1): historical perspective, phenotypes, mechanism, pathology, and epidemiology. Clin Neuropsychol. 2016 Aug;30(6):815-33. doi: 10.1080/13854046.2016.1184652. Epub 2016 Jun 29. PMID 27356167
- [Background] Wang LW, Berry-Kravis E, Hagerman RJ. Fragile X: leading the way for targeted treatments in autism. Neurotherapeutics. 2010 Jul;7(3):264-74. doi: 10.1016/j.nurt.2010.05.005. PMID 20643379
- [Background] Hagerman RJ, Berry-Kravis E, Hazlett HC, Bailey DB Jr, Moine H, Kooy RF, Tassone F, Gantois I, Sonenberg N, Mandel JL, Hagerman PJ. Fragile X syndrome. Nat Rev Dis Primers. 2017 Sep 29;3:17065. doi: 10.1038/nrdp.2017.65. PMID 28960184
- [Background] Quartier A, Poquet H, Gilbert-Dussardier B, Rossi M, Casteleyn AS, Portes VD, Feger C, Nourisson E, Kuentz P, Redin C, Thevenon J, Mosca-Boidron AL, Callier P, Muller J, Lesca G, Huet F, Geoffroy V, El Chehadeh S, Jung M, Trojak B, Le Gras S, Lehalle D, Jost B, Maury S, Masurel A, Edery P, Thauvin-Robinet C, Gerard B, Mandel JL, Faivre L, Piton A. Intragenic FMR1 disease-causing variants: a significant mutational mechanism leading to Fragile-X syndrome. Eur J Hum Genet. 2017 Apr;25(4):423-431. doi: 10.1038/ejhg.2016.204. Epub 2017 Feb 8. PMID 28176767
- [Background] Myrick LK, Nakamoto-Kinoshita M, Lindor NM, Kirmani S, Cheng X, Warren ST. Fragile X syndrome due to a missense mutation. Eur J Hum Genet. 2014 Oct;22(10):1185-9. doi: 10.1038/ejhg.2013.311. Epub 2014 Jan 22. PMID 24448548